CLINICAL TRIAL: NCT02736331
Title: The Effect of Different Types of Fruits on Metabolic Function and Cognitive Performance
Brief Title: Different Types of Fruits on Metabolic Function and Cognitive Performance
Acronym: WBB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB2015-105
Record Dates: First submitted 2016-03-31; First posted 2016-04-13 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Cognitive performance; Metabolic control; Pharmacokinetic profile; Anthocyanins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 Beverage (Experimental): Treatment 1
  Interventions: Dietary Supplement: Treatment 1
- Treatment 2 Beverage (Placebo Comparator): Treatment 2
  Interventions: Dietary Supplement: Treatment 2

INTERVENTIONS:
Dietary Supplement: Treatment 1 — Treatment 1 Beverage
  Arms: Treatment 1 Beverage
Dietary Supplement: Treatment 2 — Treatment 2 Beverage
  Arms: Treatment 2 Beverage

SUMMARY:
Primary objective is to assess the effect of the intake of different types of fruits on memory and attention.

Secondary objective is to assess effect of intake of different types of fruits on metabolic markers, including glucose, insulin, total cholesterol and triglyceride and the pharmacokinetic profile of the anthocyanins.

DETAILED DESCRIPTION:
The trial is designed as a randomized 2-arm, placebo-controlled, within-subjects crossover utilizing a multiple sampling, repeated measures paradigm to investigate the effects of consumption of different types of fruits on cognitive performance and metabolic responses. This trial will test 2 treatment conditions in forty men and women who will be enrolled into the study.

Each subject will be asked to come for one screening visit, a pre-study visit, and two dinner pick-ups the day before each of the two test visits and 2 test visits. Participation in this study will last approximately four weeks.

The initial screening visit will provide the subject with the informed consent document and determine eligibility through anthropometric measurements, vital signs, fasting blood glucose test , vein assessment, color test and completion of a survey relate to general eating, health, and exercise habits. In addition, subjects will take brief tests of attention and memory to ensure capability and willingness to perform tests during subsequent research visits. Eligible subjects will be trained and instructed to record all food and beverages consumed for a 3-day period (one weekend day and two weekdays) on food record diaries. At the pre-study visit, subjects will be instructed to follow a strictly limited polyphenolic diet for 7 days prior to the study and throughout their participation time, while maintaining their usual diet pattern and physical activity. A dinner meal will be provided the day before the study visit.

At each test visit, subjects will arrive at the clinic after fasting 8 to 12 hours and in a well-hydrated state. After confirming compliance with protocol, anthropometric measurements and vital signs will be taken along with a finger prick for fasting blood glucose and a catheter placement .

Fasting baseline blood sample from a catheter will be collected after which baseline cognitive performance measures will be assessed. After completing baseline measures, subjects will receive a standard breakfast meal along with a beverage containing different fruits according to the randomization sequence. Additional blood samples will be taken at 30, 60, 120, 180, 240, 300, 360, and 480 minutes after the start of the breakfast meal. Additional cognitive tests will be performed at the 120, 240, 360, and 480 minute time points. A standardized lunch will be provided between the 360 and 480 minute time points.

Subject will come to the clinic for 2 test day visits; all procedures will be the same except for the treatment (the test or control treatment).

ELIGIBILITY:
Inclusion Criteria:

* • Subject is male or female aged between 40 and 65 years of age

  * Subject has BMI between 18.5 and 34.9 kg/m2, (inclusive) at screening visit
  * Fasting blood sugar less than 126 mg/dL
  * Average Blood pressure less than 160/100 mmHg
  * Subject is willing to maintain a stable body weight and to follow his/her regular diet and physical activity patterns throughout the study period.
  * Subject is willing to refrain from vigorous physical activity and consumption of alcoholic and/or caffeinated beverages 24 h prior to each test day
  * Subject does not smoke or has abstained from smoking for at least 2 years
  * No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
  * Not taking any medications or dietary supplements that would interfere with outcomes of the study.

Exclusion Criteria:

* • Subject currently smokes or has smoked within the past 2 years

  * Subject works overnight i.e. the night shift
  * Subjects who have a significant sleep disorder, a traumatic brain injury, have a learning disability or attention deficit disorder or any psychiatric or neurological disturbances
  * Subject is color blind, has impaired cognitive performance on the flanker test (score <60 at screening) or has a vein access score <7
  * Men and women with known or suspected food intolerance, allergies or hypersensitivity to the study materials or closely related compounds
  * Men and women known to have/diagnosed with diabetes mellitus
  * Men and women with a fasting blood glucose concentration ≥126 mg/dL
  * Average blood pressure > 160/100 mmHg during screening visit
  * Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries
  * Men and women with cancer other than non-melanoma skin cancer in previous 2 years
  * Men and women who are taking medication or dietary supplements that may interfere with the study procedures or the endpoints of the study (e.g. antioxidants, anti-inflammatory medications, antidepressant medications, oral and injectable hypoglycemic medications, GI medications, antibiotics, diuretics, adrenergic blockers etc.) Subjects may choose to go off dietary supplements (requires 30 days washout)
  * Men and women taking antibiotics within 5 days of study start
  * Men and women who have donated blood/plasma within 3 months of the screening visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months
  * Substance (alcohol or drug) abuse within the last 2 years
  * Excessive coffee and tea consumption (> 4 cups/day)
  * Unstable body weight fluctuations of >4.5kg (9.9lbs) in the past 4 weeks
  * Women who are known to be pregnant or who are intending to become pregnant over the course of the study and women who are lactating.
  * Men and women whom investigator is uncertain about subject's capability or willingness to comply with protocol requirements
  * Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months.
  * Men and women who do excessive exercise regularly or are athlete

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in memory function using the Montreal Cognitive Assessment after intake of different types of fruits | 8 hours Postprandial Study
  Sum all sub-scores of the Montreal Cognitive Assessment

SECONDARY OUTCOMES:
Changes in plasma glucose concentrations after intake of different types of fruits | 8 hours Postprandial Study
  plasma glucose concentrations after intake of different types of fruits
Changes in plasma insulin concentrations after intake of different types of fruits | 8 hours Postprandial Study
  insulin concentrations after intake of different types of fruits
Changes in plasma Triglycerides Concentrations after intake of different types of fruits | 8 hours Postprandial Study
  Plasma Triglycerides Concentrations after intake of different types of fruits
Changes in plasma Total Cholesterol Concentrations after intake of different types of fruits | 8 hours Postprandial Study
  plasma Total Cholesterol Concentrations after intake of different types of fruits

OTHER OUTCOMES:
Changes in polyphenol anthocyanin concentrations after intake of different types of fruits | 8 hours Postprandial Study
  polyphenol anthocyanin concentrations after intake of different types of fruits
Changes in LDL oxidation after intake of different types of fruits | 8 hours Postprandial Study
  OxLDL after intake of different types of fruits
Changes in IL-6 after intake of different types of fruits | 8 hours Postprandial Study
  IL-6 after intake of different types of fruits
Changes in IL-1beta after intake of different types of fruits | 8 hours Postprandial Study
  IL-1beta after intake of different types of fruits
Changes in IL-10 after intake of different types of fruits | 8 hours Postprandial Study
  IL-10 after intake of different types of fruits
Changes in MCP-1 after intake of different types of fruits | 8 hours Postprandial Study
  MCP-1 after intake of different types of fruits

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No